CLINICAL TRIAL: NCT03601949
Title: A Prospective, Multi-center, Randomized, Assessor Blind, Controlled Study Comparing Lateral Branch Cooled Radiofrequency Denervation to Conservative Therapy as Treatment for Sacroiliac Joint Pain in a Military and Civilian Population
Brief Title: Lateral Branch Cooled Radiofrequency Denervation vs. Conservative Therapy for Sacroiliac Joint Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Avanos Medical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 105-17-0002
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Sacroiliac Joint Pain
Keywords: Back Pain; Low Back Pain; Sacroiliac Back Pain
MeSH Terms: conditions — Back Pain; Low Back Pain | interventions — Practice Management, Medical

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study is an assessor blinded trial and deliberate action will be needed to ensure the blind remains. This begins with randomization procedures and carries through the follow up visits. It is suggested that all follow up visit documentation not contain the visit number, but instead utilize visit dates to track progress.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- SInergy Cooled Radiofrequency (Experimental): Halyard Health SInergy Cooled Radiofrequency in addition to standard medical management
  Interventions: Device: SInergy Cooled Radiofrequency; Other: Medical Management
- Medical Management (Active Comparator): Standard Medical Management
  Interventions: Other: Medical Management

INTERVENTIONS:
Device: SInergy Cooled Radiofrequency — ablation of low back pain
  Other Names: SInergy
  Arms: SInergy Cooled Radiofrequency
Other: Medical Management — physical therapy, medications, lifestyle changes
  Other Names: Standard Medical Management

SUMMARY:
This is a prospective, randomized, controlled, multi-center clinical study. Approximately 208 subjects will be enrolled at approximately 12-15 active duty military, veterans' care, and civilian sites. Eligible subjects will be randomized in 1:1 ratio to receive either Sacroiliac denervation using CRF (treatment group) or standard medical management ("SMM," control group).

DETAILED DESCRIPTION:
This study will be a 12-month prospective, randomized, controlled, prospective, open-label, multi-center clinical study. Adult subjects over the age of 21 with diagnosed chronic intractable sacroiliac joint pain (≥ 3 months), who have been previously unresponsive to conservative therapy and who meet the selection criteria are eligible to participate in this study. Approximately 208 subjects will be enrolled at up to 15 sites in a 1:1 randomization ratio to receive either denervation using the SInergy System (cooled radiofrequency (CRF), treatment group) or standard medical management (SMM, control group). Follow-up will be conducted for a total of 12 months post-Coolief (cooled radiofrequency ablation) procedure, with the primary endpoint being completed at month 3. The control arm will utilize physician prescribed standard medical management (SMM). For this protocol, this includes, but is not limited to, medications, physical therapy, lifestyle changes, acupuncture, yoga, chiropractic, and therapeutic injections. An optional crossover-to-treatment design was adopted for subjects randomized to standard medical management after their 3-month visit, because it would be considered unethical to withhold treatment that could potentially offer pain relief to those subjects undergoing standard medical management who continue to suffer from pain.

Eligibility includes BOTH of the following:

* 50% pain relief lasting for the expected duration of anesthetic or medication from a therapeutic or diagnostic sacroiliac joint injection; AND

  * 50% pain relief lasting for the expected duration of anesthetic from a standardized set of lateral branch blocks, with total volume of no more than 1 milliliter (ml) of 0.5% Bupivacaine, Ropivacaine (or similar). Ideally, 0.5 ml will be utilized at L5 and the remaining 0.5 ml should be divided in at least two locations along the foramen line

After the CRF treatment, the CRF treatment group subjects will visit the blinded assessor for follow up at 1, 3, 6, 9, and 12 months. At the month 3 visit (three months post-randomization), subjects initially randomized to the conservative therapy group will be assessed to determine eligibility to receive CRF treatment.

* If the conservative treatment subjects fail conservative therapy at 3 months (defined as failure to obtain a 2-point decrease in average pain score from baseline AND failure to obtain a rating of at least 5 on the Patient Global Impression of Change (PGIC) scale), they will be given the option of receiving CRF treatment.
* Subjects who choose to cross-over will ideally receive treatment within 30 days of their 3-month visit but they must receive treatment within 90 days of their 3-month visit. They will then be followed-up at 1, 3, 6, 9, and 12 months following CRF denervation (new Day 0).
* If the conservative treatment group subjects refuse or don't qualify for CRF treatment at 3 months, they will subsequently be followed-up at 6, 9, and 12 months from their Day 0.

Primary Analysis is planned after all initially treated subjects have completed their 3-month post-procedure visit.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 21 years.
2. Able to understand the informed consent, and able to complete outcome measures.
3. Sacroiliac joint (SIJ) pain that is refractory to standard of care treatments such as non-steroidal anti-inflammatory drugs (NSAIDS), physical therapy, etc.
4. At least one positive SIJ pain provocation test (Distraction, Gaenslen's, FABER, Sacral Sulcus tenderness, thigh thrust, compression or sacral thrust).
5. Back pain is predominantly below the lumbar (L) 5 vertebrae.
6. Chronic low back pain lasting for longer than three months.
7. Greater than 50% pain relief lasting for the expected duration of anesthetic or medication from a therapeutic or diagnostic SIJ injection.
8. Greater than 50% pain relief lasting the duration of anesthetic from lateral branch block (done on different days than SIJ injection).
9. Stabilized on pain medication regimen for > 2 months, as defined by a < 10% change in dosage.
10. Numeric rating scale indicating an average pain score of > 4 over the last seven days. (returned to pre-lateral branch block baseline pain).
11. All other possible sources of low back pain have been ruled out as the primary pain generator, including, but not limited to: suspected advanced degenerative joint disease, the intervertebral discs, bone fracture, the zygapophyseal joints, the hip joint, symptomatic spondylolisthesis, tumor, and other regional soft tissue structures (this is done by physical exam, medical history, and magnetic resonance imaging/computed tomography/X-ray, as required).
12. Willing to utilize double barrier contraceptive method, if of child-bearing potential.
13. Willingness to provide informed consent and to comply with the requirements of this protocol for the full duration of the study.
14. Physician believes ablation of the SIJ is an appropriate treatment for the patient.

Exclusion Criteria:

1. Poorly controlled severe psychiatric illness or ongoing psychological barriers to recovery, as determined by the treating physician.
2. Spinal pathology that may impede recovery such as spina bifida occulta, grade II or higher spondylolisthesis at vertebrae L5/sacroiliac (S) 1, or scoliosis.
3. Symptomatic moderate or severe foraminal or central canal stenosis.
4. Systemic infection or localized infection at anticipated introducer entry site.
5. Uncontrolled immunosuppression (e.g., acquired immune deficiency syndrome (AIDS), cancer, diabetes, etc.)
6. Chronic severe conditions such as rheumatoid/inflammatory arthritis.
7. Pregnancy or recent delivery (within three months).
8. Active radiculopathy pain from lumbar spine.
9. Active hip pathology.
10. Major surgery within three months prior to signing informed consent.
11. Prior radiofrequency denervation of the lateral sacral nerves.
12. Ongoing/unresolved worker's compensation, injury litigation, military medical board, or disability remuneration claims.
13. Allergy to injected substances or medications used in procedure.
14. Body mass index (BMI) > 40 kilograms/meter (squared).
15. Current prescribed opioid medications equivalent to 90 mg of morphine per 24 hours or greater.
16. Subject is currently implanted with pacemaker, stimulator, or defibrillator.
17. Participation in another clinical trial/investigation that could interfere with this trial 30 days prior to signing informed consent.
18. Subject is unwilling or unable to comply with the protocol requirements.

Ages: 21 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2018-06-29 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2022-06-23 (Actual)

PRIMARY OUTCOMES:
Change in average daily pain Numeric Rating Scale (NRS) score | Baseline and 3 months
  Numeric Rating Scale (NRS) - score range = 0 - 10. "0" corresponds to "no pain" and "10" indicates "worst pain imaginable". The means of these scores and their respective standard deviations are reported for each study group.

SECONDARY OUTCOMES:
The proportion of subjects with at least a 2 points decrease or 30% drop in average daily pain related NRS score AND a rating of at least 5 on the Patient Global Impression of Change (PGIC) | Baseline and 3 months
  Numeric Rating Scale (NRS) - score range = 0 - 10. "0" corresponds to "no pain" and "10" indicates "worst pain imaginable". The means of these scores and their respective standard deviations are reported for each study group. PGIC - score range = 1 - 7. "1" corresponds to "very much improved" and "7" indicates "very much worse" pertaining to overall activity, symptoms, emotions, and quality of life. The means of these scores and their respective standard deviations are reported for each study group.
Mean change in score of Patient Global Impression of Change (PGIC) | Baseline and 3 months
  PGIC - score range = 1 - 7. "1" corresponds to "very much improved" and "7" indicates "very much worse" pertaining to overall activity, symptoms, emotions, and quality of life. The means of these scores and their respective standard deviations are reported for each study group.
Mean change in score of Short Form 36-Physical Functioning (SF36-PF) | Baseline and 3 months
  Short Form 36-PF - score range = 0 - 100. "0" corresponds to "greatest disability" and "100" indicates "no disability". The means of these scores and their respective standard deviations are reported for each study group.
Mean change in score of Oswestry Disability Index (ODI) | Baseline and 3 months
  ODI - score range = 0 - 100. "0" corresponds to "no disability" and "100" indicates the "maximum disability possible". The means of these scores and their respective standard deviations are reported for each study group.
Mean change in score of EuroQuol (EQ) 5D-5L | Baseline and 3 months
  This tool involves two components: 1) descriptive system - five questions that are scored 1-5, each with "1" indicating no problems and "5" indicating the worst problem related to the question, and 2) EQ-Visual Analog Scale (VAS) - score range = 0 - 100. "0" corresponds to the "worst imaginable health state" and "100" indicates the "best imaginable health state". The means of these scores and their respective standard deviations are reported for each study group.

OTHER OUTCOMES:
The mean change in pain-related medication | Baseline and 3 months
  The absolute mean difference between analgesic use at baseline and that at 3 months post-randomization.
Healthcare Utilization Questionnaire | Baseline and 3 months
  Used to evaluate the use or need for other healthcare treatments (e.g., physical therapy, visit(s) to chiropractor). The evaluation is not based on a point-based scale, but rather is based on responses made by trial subjects to the questions, with the determination made by the investigator.
Time from treatment to return to work/duty | 3 months post-intervention
  Trial subject will be asked if/when she/he returned to work/duty
Time from treatment to return of pain date | 3 months post-intervention
  Trial subject will be asked if/when she/he experienced a return of pain

CONTACTS AND LOCATIONS:
Overall Officials: David Curd, MS, Study Director — Avanos Medical
Locations (15):
- United States (15):
  - Mehul Desai, Washington D.C., District of Columbia
  - Millennium Pain Center, Bloomington, Illinois
  - Ochsner Medical Center, New Orleans, Louisiana
  - Shravani Durbhakula, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Brigham and Women's Hospital, Chestnut Hill, Massachusetts
  - Premier Pain Centers, Shrewsbury, New Jersey
  - Adam Carinci, Rochester, New York
  - Womack Army Medical Center, Fort Bragg, North Carolina
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - Clinical Investigations, Edmond, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Lynn Kohan, Charlottesville, Virginia
  - Michael DePalma, Richmond, Virginia

REFERENCES:
- [Derived] Cohen SP, Kapural L, Kohan L, Li S, Hurley R, Vallejo R, Eshraghi Y, Dinakar P, Durbhakula S, Beall DP, Desai MJ, Reece D, Christiansen S, Chang MH, Carinci AJ, DePalma M. Cooled radiofrequency ablation provides extended clinical utility in the management of chronic sacroiliac joint pain: 12-month follow-up results from the observational phase of a randomized, multicenter, comparative-effectiveness crossover study. Reg Anesth Pain Med. 2025 Mar 15:rapm-2024-106315. doi: 10.1136/rapm-2024-106315. Online ahead of print. PMID 40089310
- [Derived] Cohen SP, Kapural L, Kohan L, Li S, Hurley RW, Vallejo R, Eshraghi Y, Dinakar P, Durbhakula S, Beall DP, Desai MJ, Reece D, Christiansen S, Chang MH, Carinci AJ, DePalma M. Cooled radiofrequency ablation versus standard medical management for chronic sacroiliac joint pain: a multicenter, randomized comparative effectiveness study. Reg Anesth Pain Med. 2024 Mar 4;49(3):184-191. doi: 10.1136/rapm-2023-104568. PMID 37407279